CLINICAL TRIAL: NCT02220205
Title: Evaluation of the PelvicSim Simulator for Training in Intrauterine Device Insertions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Siripanth Nippita, Instructor in Obstetrics, Gynecology and Reproductive Biology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2014P-000106
Record Dates: First submitted 2014-08-14; First posted 2014-08-19 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-04

CONDITIONS: Contraceptive Devices, Intrauterine; Education, Medical
Keywords: IUD; training; simulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PelvicSim (Active Comparator): Participants randomized to this arm practice IUD insertion on the PelvicSim for 30 minutes.
  Interventions: Other: PelvicSim
- Manufacturer model (Placebo Comparator): Participants randomized to this arm practice IUD insertion on models provided by the IUD manufacturer for 30 minutes.
  Interventions: Device: Manufacturer model

INTERVENTIONS:
Other: PelvicSim
  Arms: PelvicSim
Device: Manufacturer model
  Arms: Manufacturer model

SUMMARY:
Intrauterine devices (IUDs) are a very effective, long-acting method of contraception. In order to make them accessible to women, health care providers must be trained to insert them. Physicians, physician assistant, and nurse practitioners often learn how to do so by first learning about IUDs, then practicing on a model that the IUD manufacturer provides.

Educators have recently been using more sophisticated models to teach clinical skills such as surgical procedures. We are investigating whether these models may be more useful in teaching IUD insertion.

ELIGIBILITY:
Inclusion Criteria:

* First-year residents in obstetrics and gynecology or family medicine, or student in physician assistant or nurse practitioner training programs
* Trainees who have performed <5 intrauterine device insertions
* Trainees who plan to provide intrauterine devices in their clinical practice

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Siripanth Nippita, MD, MS, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant voluntarily withdrew from the study due to time constraints which precluded completion of the study visit. Therefore, 60 participants enrolled and were randomized, and 59 completed the study.
Groups:
- PelvicSim: Participants randomized to this arm practice IUD insertion on the PelvicSim for 30 minutes.
  PelvicSim
- Manufacturer Model: Participants randomized to this arm practice IUD insertion on models provided by the IUD manufacturer for 30 minutes.
  Manufacturer model
Period: Overall Study
Arm/Group | PelvicSim | Manufacturer Model
Started | 30 | 30
Completed | 29 | 30
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PelvicSim | Manufacturer Model | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 26 [26 to 30] | 28 [26 to 30] | 27 [26 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 26 | 53
  Male | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 29 | 30 | 59
Occupation [Number; unit: participants] — Intern or NP student
  participants
    Intern | 8 | 12 | 20
    Nurse practitioner student | 21 | 18 | 39
Prior pelvic exams [Number; unit: exams]
  0 | 10 | 5 | 15
  1-5 | 10 | 10 | 20
  6-10 | 2 | 6 | 8
  >10 | 7 | 9 | 16
Prior IUD insertions performed [Number; unit: exams]
  >=1 | 6 | 2 | 8
  0 | 23 | 28 | 51

OUTCOME MEASURES:

1. Primary Outcome: Insertion Score Before and Immediately After Initial Practice (Same Day), and 3 Months After Initial Practice
Description: Participants were filmed performing 3 IUD insertions each, for three IUDs available in the US. They then practiced on an assigned simulator for 30 minutes, and were re-recorded immediately afterwards. Three months after initial practice, they returned and performed the insertions again.
  Sets of insertions were scored using a checklist. Participants earned up to 86 points for performing various elements of IUC insertion correctly: sounding the uterus (14 points), and loading as well as inserting the copper device (24 points), levonorgestrel 52mg device (26 points), and levonorgestrel 13.5mg device (22 points). Higher scores were better.
Time Frame: Before and immediately after initial practice on assigned simulator (same day), and three months after initial practice
Measure: Median (Inter-Quartile Range); unit: Percent of tasks performed correctly
Arm/Group | PelvicSim | Manufacturer Model
Number analyzed (Participants) | 29 | 30
Percent of tasks performed correctly
  Pre-simulation | 61.5 [50 to 69] | 67.5 [53 to 76]
  Post-simulation | 82.5 [72 to 88] | 83 [73 to 91]
  Three month visit | 65.5 [58 to 75] | 67.5 [59 to 76]

2. Secondary Outcome: Percent Change in Comfort Placing IUDs From Pre- to Post-insertion
Description: Participants were given questionnaires at the initial study visit and at a three-month follow-up visit that assessed their comfort with IUD insertion using a modified Likert scale.
Time Frame: Baseline to three months
Measure: Number; unit: Percent change in comfort
Arm/Group | PelvicSim | Manufacturer Model
Number analyzed (Participants) | 29 | 30
Percent change in comfort
  Copper IUD | 89.3 | 96.7
  52mg levonorgestrel IUD | 92.9 | 100
  13.5mg levonorgestrel IUD | 89.3 | 100

ADVERSE EVENTS:
Arm/Group | PelvicSim | Manufacturer Model
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 0/29 | 0/30

LIMITATIONS AND CAVEATS:
Participants directed their own practice time. An investigator answered questions but did not provide other feedback unless specifically asked.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No